CLINICAL TRIAL: NCT04804358
Title: Study of the Difference Between Anorexia Nervosa with a History (s) of Psychological Trauma (AM-T) and Classical Anorexia Nervosa (AM-C) on the Neurocognitive and Neurophysiological Factors
Brief Title: Study of the Difference Between Anorexia Nervosa with a History of Psychological Trauma and Classical Anorexia Nervosa on the Neurocognitive and Neurophysiological Factors
Acronym: ATAC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The person in charge of the clinical study had to leave the hospital prematurely.
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RECHMPL20_0186
Record Dates: First submitted 2021-03-10; First posted 2021-03-18 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; Psychological Trauma; Heart Rate Variability; Kynurenine; Substance P
MeSH Terms: conditions — Anorexia Nervosa; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Anorexic women (Other): Anorexic women with or without history of psychological trauma will perform study procedure : sociodemographic and clinical assessments, measurement of cardiac variability and salivary cortisol changes, before, during and after the exposition test.
  Interventions: Behavioral: Exposition Test

INTERVENTIONS:
Behavioral: Exposition Test — During this test (7 minutes) participants will be exposed to photos evoking positive or negative emotions (anger, disgust, sadness and fear) interspersed with emotionally neutral photos.
  The test sequence is composed of 3 blocks as follows:
  * 12 photos evoking positive emotions (2 min)
  * Pause of 30 seconds (white screen)
  * 12 photos presenting a neutral emotional valence (2 min)
  * Pause of 30 seconds (white screen)
  * 12 photos evoking negative emotions (2min)
  In each block, photos will be selected and presented to the participant in a randomized and sequential manner. In total, 30 photos will be presented in 7 minutes to each participant (10 seconds per photo).
  The participant must be at rest in front of the computer screen during these 7 minutes with optimal visibility. The photos will be presented sequentially using software (E-Prime or Visual Basic 6.0). During this exposure test, a heart rate recording will be made using a BIOPAC MP160 recording system.

SUMMARY:
Recent studies suggest that patients with an history of trauma may represent a specific subtype of anorexia nervosa (AM) underlined by specific neurobiological and psychopathological mechanisms. Thus, AM-T subjects would manifest cognitive (specific difficulties in executive functions), emotional (emotional disruption, impulsivity, etc.) and neurobiological (secretion of kynurenine and neurokinins in the face of stress) caracteristics different from those of AM subjects.

DETAILED DESCRIPTION:
We will recruit a total of 100 patients with a diagnosis of anorexia nervosa in the university hospital of Montpellier : 50 patients with an history of psychological trauma and 50 patients without any history of psychological trauma

Participation consists of a half-day visit. Patients will perform clinical and neuropsychological assessments and an exposition test. During this test, participants will be exposed, for 7 minutes, to neutral, positive or negative emotional photos. Heart rate variability will be determined through a Biopac MP160 before, during and after this event. Saliva samples to measure kynurenin, tryptophan, substance P and neurokinin-1 will be collected before and directly after the test.

ELIGIBILITY:
Inclusion criteria common to the 2 groups AM-T and AM-C :

* Women Patient
* Present a diagnosis of anorexia nervosa according to the DSM-5 criteria
* Between 18 and 65 years old
* Present a BMI> 14
* Do not present a sight problem or be corrected appropriately by wearing glasses or contact lenses.
* Be affiliated to a social security scheme, or beneficiary of such a scheme
* Be able to understand the nature, purpose and methodology of the study

Inclusion criteria specific to patients in the AM-T group:

- To have answered at least one of the grayed out items of the LEC-5, that is to say to have answered "it happened to me" to at least one of the items 1 to 13 or to item 16 "and / or having answered" I witnessed it "to at least one of items 14 and 15.

Inclusion criteria specific to patients in the AM-C group:

- Not having answered "it happened to me" or "I witnessed it" to one of the items of LEC-5

Exclusion Criteria:

* Present a severe unstable mental pathology in the opinion of the investigator
* Present active suicidal ideation
* Have consumed psychoactive substances in the last 24 hours before the assessment
* Present a severe major depressive episode incompatible with the assessment, in the opinion of the investigator.
* Present in the opinion of the investigator an unstable somatic state (eg severe metabolic disorder making it impossible or likely to impair the reliability of neuropsychological and cardiac evaluations).
* Take a drug treatment acting on the cardiovascular system
* Refusal of the patient
* Be protected by law (tutorship or curatorship).
* To be deprived of liberty by administrative decision.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Changes in high frequency heart variability (HF-HRV) across the exposition test (before, during and after) | inclusion visit
  We aim to investigate if AM-T patients present changes in HF-HRV across exposition test compared to AM-C patients, measured by Biopac MP160

SECONDARY OUTCOMES:
Changes in low frequency heart variability (LF-HRV) across the exposition test (before, during and after) | inclusion visit
  We aim to investigate if AM-T patients present changes in LF-HRV across exposition test compared to AM-C patients, measured by Biopac MP160
Changes in very low frequency heart variability (VLF-HRV) across the exposition test (before, during and after) | inclusion visit
  We aim to investigate if AM-T patients present changes in VLF-HRV across exposition test compared to AM-C patients, measured by Biopac MP160
Changes in the highest peak of the high frequency (HFhz) across the exposition test (before, during and after) | inclusion visit
  We aim to investigate if AM-T patients present changes in HFhz across exposition test compared to AM-C patients, measured by Biopac MP160
Changes in the interval between R peaks (R-R across the exposition test (before, during and after) | inclusion visit
  We aim to investigate if AM-T patients present R-R changes across exposition test compared to AM-C patients, measured by Biopac MP160
Changes in the R-R interval standard difference (STD-RR) across the exposition test (before, during and after) | inclusion visit
  We aim to investigate if AM-T patients present STD-RR changes across exposition test compared to AM-C patients, measured by Biopac MP160
Changes in the root mean successive squared differences of the R-R interval (RMSSD). across the exposition test (before, during and after) | inclusion visit
  We aim to investigate if AM-T patients present RMSSD changes across exposition test compared to AM-C patients, measured by Biopac MP160
Score to the Difficulties in Emotion Regulation Scale | inclusion visit
  We aim to assess the link between emotional regulation and psychological trauma in AN. DERS is a self-assessment scale measuring emotion dysregulation. The original DERS includes 36 items scored 1-5 where 1 is almost never, 2 is sometimes, 3 is about half the time, 4 is most of the time, and 5 is almost always. Of the 36 items, 11 are reverse scored. The DERS-36 yields a total score as well as six subscales where higher scores indicate more difficulties.
Score to the Beck depression inventory II | inclusion visit
  We aim to assess the link between eating symptomatology and psychological trauma in AN. The BDI-II is a self-administered questionnaire assessing the severity of depressive symptoms in 21 items. Each item is rated on a 4-points Likert scale ranging from 0 to 3. The total score varies between 0 and 63. higher scores mean more depressive symptoms
Score to the Eating Disorder Questionnaire | inclusion visit
  We aim to assess the link betxeen eating symptomatology and psychological trauma in AN. self-administered questionnaire assessing the intensity of eating symptoms over the past 28 days. A total score as well as 4 sub-scores (restriction, diet, weight, shape) varying from 0 to 6 are obtained.Higher scores mean higher eating concerns
Score to the Eating Disorder Inventory | inclusion visit
  We aim to assess the link between eating symptomatology and psychological trauma in AN. The EDI-2 is a 91-item self-report questionnaire assessing cognitive, emotional, and behavioral symptoms of eating disorders. It rates from 0 to 273. Higher scores means severe symptoms
Score to the Childhood trauma questionnaire | inclusion visit
Score to the PTSD Checklist for DSM-5 | inclusion visit
Score to the Wisconson Card Sorting Test | inclusion visit
  We aim to assess the link between mental flexibility, working memory, inhibition and psychological trauma in AN
Score to the Stroop Test | inclusion visit
  We aim to assess the link between mental flexibility, working memory, inhibition and psychological trauma in AN
Score to the Delay Discounting Test | inclusion visit
  We aim to assess the link between decision making and psychological trauma in AN
Score to the Trail Making Test | inclusion visit
  We aim to assess the link between mental flexibility, visio-spatial attention, processing speed and psychological trauma in AN
Changes in salivary tryptophan | inclusion visit
  study changes in salivary tryptophan before and after exposition test
Changes in salivary kynurenine | inclusion visit
  study changes in salivary kynurenine before and after exposition test
Changes in salivary P substance | inclusion visit
  study changes in salivary P substance before and after exposition test
Changes in salivary neurokinin-1 | inclusion visit
  study changes in salivary neurokinin-1before and after exposition test

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Montpellier, Montpellier, France